CLINICAL TRIAL: NCT06710808
Title: VIRTUAL WALKING AND TRANSCRANIAL DIRECT CURRENT STIMULATION (TDCS) FOR CHRONIC NEUROPATHIC PAIN DUE TO SPINAL CORD INJURY (SCI): A FEASIBILITY STUDY
Brief Title: VIRTUAL WALKING AND TRANSCRANIAL DIRECT CURRENT STIMULATION FOR CHRONIC NEUROPATHIC PAIN DUE TO SPINAL CORD INJURY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-12
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury; Chronic Neuropathic Pain
Keywords: Neuropathic pain; Chronic neuropathic pain; spinal cord injury; virtual walking; transcranial direct current stimulation; tDCS
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual walking and transcranial direct current stimulation of 2 milliampere for 20 minutes (Experimental)
  Interventions: Other: Virtual walking and transcranial direct current stimulation

INTERVENTIONS:
Other: Virtual walking and transcranial direct current stimulation — Participants will receive VW-therapy combined with tDCS. The intervention is adapted from Soler et al. 2010 and consists of 10 sessions over 2 weeks, each session lasting around 20 minutes.
  For the virtual walking the participant sits on a modified wheelchair, which is positioned at a distance of two meters from the screen. The setting provides an illusion of a third person perspective and the participant can see himself/herself walk through a forest ambience.
  The tDCS session is according the same protocol from Soler et al., 2010. Hereby, the device from Starstim, Neuroelectrics will be used, which is equipped with a neoprene cap containing electrodes. The anodes will be placed over C3 or C4 (EEG 10/20 system) to target the motor cortex (M1) contralateral to the painful side and the cathodes will be placed over the contralateral supraorbital area. Symmetric pain participants receive stimulation on the dominant hemisphere. The tDCS applies a constant current of 2 mA over 20 minutes.

SUMMARY:
The goal of this feasibility study is to assess the feasibility of the combined treatment intervention "virtual walking (VW) and transcranial direct current stimulation (tDCS)" of neuropathic pain in patients with spinal cord injury. The main question aims to answer:

• To assess the feasibility of combining VW and tDCS for longer-term use from the patients' point of view.

Participants will:

Receive a two week intervention in the Swiss Paraplegic Centre in Nottwil, where the participants undergo VW and tDCS for ten sessions, each lasting around 20 minutes.

The participants keep a diary and a pain drawing of their symptoms and will fill out some questionnaires about their impression of feasibility, the pain intensity, chronicity, the impression of change, depression, anxiety, stress and adverse events. At the beginning and end of the study the participants will be interviewed about their expectations, hopes and the feasibility of the procedures from a participants point of view.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18y, ≤ 75y
* traumatic SCI (> 6 month after SCI) with a SCI severity grade AIS A, B, C or D
* At or below level spinal cord injury neuropathic pain on trunk or lower extremities according to the ISCIP classification (Bryce et al., 2012) of at least 4/10 intensity on a NRS (Langford et al., 2023) with in the last 7 days (WiderströmNoga et al., 2023)
* Good communication in German to understand the instructions, assessments and to fill in questionnaires
* Adequate siting balance
* Ability to draw with a pencil
* Ability to swing arms

Exclusion Criteria:

* severe psychiatric disorder requiring psychiatric hospitalisation or mental disease that could interfere with their ability to participate
* Previous brain surgery
* Metal implants in the skull or brain, including cochlear implants, intracranial electrodes or a pacemaker (Datta et al., 2010)
* Drugs that affect cortical excitability (McLaren et al., 2018): Alcohol, Amphetamines, Theophylline (asthma treatment), Chlorpromazine, Clozapine, Amitriptyline, Doxepine, Imipramine, Maprotiline, Nortriptyline, Foscarnet, Ganciclovir, Ritonavir, Amphetamines, Cocaine, Gamma-hydroxybutyrate (GHB), Ketamine, MDMA, ecstasy Phencyclidine
* Previous adverse effects of stimulation with tDCS
* A scalp or skin condition (e.g. psoriasis or eczema)
* History of epilepsy or seizure
* Pregnancy (anamnestic)
* Inability to give consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Patient-reported expectations, acceptability and satisfaction | one week before treatment, 2 weeks during treatment, 1 week after treatment
  semistructured interview

SECONDARY OUTCOMES:
Adherence rate | during 2 weeks treatment
Drop out rate | during 2 weeks treatment
Preparation time | during 2 weeks treatment
  Time for preparation of participant in minutes
Quality of pain | one week pre-treatment, one week post-treatment
  Neuropathic Pain Symptom Inventory (NPSI)
Pain distribution | From enrollment to the end of study at 4 weeks
  size of the drawn area in pixels and percentage in relation to the total body chart indicated by patient into a pain drawing scheme
Pain intensity | Daily from enrollment to the end of study at 4 weeks
  Numeric Rating Scale (no pain to most imaginable pain)
Patient Global Impression of Change (PGIC) | one week post-treatment
  Subjective global impression of change after treatment
Depression, anxiety and stress | one week pre-treatment and one week post-treatment
  Depression Anxiety & Stress Scale (DASS)
Pain chronicity | one week pre-treatment
  Mainz Pain Staging System (MPSS)
Safety of tDCS | every day during the 2 weeks treatment
  Adverse events questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Switzerland

IPD SHARING:
Plan to Share IPD: No